CLINICAL TRIAL: NCT07127211
Title: Angle-Specific Upper and Lower Body Muscle Activation in Suspension Push-Ups: An Electromyographic Analysis Across Different Body Angles
Brief Title: Angle-Specific Upper and Lower Body Muscle Activation in Suspension Training
Status: Completed | Type: Observational
Sponsor: TSUNG-LIN CHIANG (Other)
Responsible Party: Sponsor-Investigator, TSUNG-LIN CHIANG, Researcher, Chinese Culture University
Organization: Chinese Culture University (Other)
Other Study IDs: No. 10711HS080
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: Suspension Training; Muscle Activation; Angle-Specific Training; unstable training; strength training
MeSH Terms: interventions — Suspensions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Suspension and Stable Push-Up Training at Multiple Angles — Participants will perform push-ups under three suspension conditions: (1) no suspension (hands and feet on a stable surface), (2) hands suspended using TRX straps, and (3) feet suspended using TRX straps. Each condition will be performed at five different body angles relative to the floor: +30°, +15°, 0°, -15°, and -30° (0° defined as shoulder joints aligned with ankle joints when arms are extended).
  For each angle, participants will complete five repetitions, with 3-5 minutes of rest between angles and at least 48 hours of rest between suspension conditions to minimize fatigue effects. All exercises will be conducted under supervision to ensure correct form and safety.
  Surface electromyography (EMG) will record muscle activity from the pectoralis major, anterior deltoid, triceps brachii, upper trapezius, and serratus anterior. EMG data will be processed as root mean square (RMS) and normalized to maximal voluntary isometric contraction (%MVIC).
  This intervention is designed to dete

SUMMARY:
The study aims to compare differences in muscle activation during push-ups performed at five body angles using different suspension methods. The investigators will recruit 20 healthy men with resistance-training experience. Each participant will perform push-ups under three suspension conditions (no suspension, hands suspended, and feet suspended) at +30°, +15°, 0°, -15°, and -30°. For each angle, participants will complete five repetitions with 3-5 minutes of rest between angles; at least 48 hours will separate suspension conditions. Surface electromyography (EMG) will record activity of the pectoralis major, anterior deltoid, triceps brachii, upper trapezius, and serratus anterior. EMG amplitudes will be normalized to maximal voluntary isometric contraction (%MVIC). Data will be analyzed using a repeated-measures two-way ANOVA to test the effects of suspension type and angle on muscle activation. The a priori hypothesis is that feet-suspended push-ups will elicit greater activation than other conditions, and that lower body angles will be associated with higher activation levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adults with ≥3 months of regular resistance-training experience.
* Able to independently perform a standard push-up with proper form.
* Willing to follow pre-session restrictions (e.g., avoid strenuous exercise within 24 h) and provide written informed consent.

Exclusion Criteria:

* Physician-diagnosed cardiovascular disease, musculoskeletal disorders, chronic pulmonary disease, or arthritis.
* Major surgery or severe injury within the past 12 months that affects physical activity.
* Current pain, injury, or functional limitation of the upper or lower limbs or trunk that would interfere with push-up performance.
* Any medical condition judged by the investigators to make participation unsafe.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy male adults with at least 3 months of regular resistance-training experience, capable of independently performing a standard push-up with proper form. Participants will be recruited from university sports facilities and local fitness centers through flyers, online announcements, and word of mouth.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Muscle Activation (%MVIC) of Upper Body Muscles During Suspension and Stable Push-Ups at Different Angles | Baseline measurement during each exercise condition within 4 weeks of study start
  Surface electromyography (EMG) will measure the root mean square (RMS) activity of the pectoralis major, anterior deltoid, triceps brachii, upper trapezius, and serratus anterior during push-ups performed under three suspension conditions (no suspension, hands suspended, feet suspended) at five body angles (+30°, +15°, 0°, -15°, -30°). RMS values will be normalized to maximal voluntary isometric contraction (%MVIC). Comparisons will be made using repeated-measures two-way ANOVA to determine the effects of suspension condition and angle on muscle activation.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Culture University, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No